CLINICAL TRIAL: NCT00526903
Title: Recurrent Abdominal Pain in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Robert Shulman, M.D., Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 17388; R01NR005337 (NIH)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Pain; Irritable Bowel Syndrome
Keywords: IBS; abdominal pain; recurrent abdominal pain; irritable bowel syndrome; diarrhea; constipation; bloating
MeSH Terms: conditions — Abdominal Pain; Irritable Bowel Syndrome; Diarrhea; Constipation | interventions — Elimination Diets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fiber (Experimental): Fiber added to diet for a total of 6 weeks.
  Interventions: Behavioral: Elimination Diet
- Placebo (Placebo Comparator): Placebo powder taken for a total of 6 weeks.
  Interventions: Behavioral: Elimination Diet

INTERVENTIONS:
Behavioral: Elimination Diet — Daily diet change for 8 days.

SUMMARY:
The purpose of this study is to:

1. To determine if fiber versus placebo improves symptoms in children with recurrent abdominal pain/irritable bowel syndrome.
2. To determine possible ways fiber or placebo improve(s) symptoms in children with recurrent abdominal pain/irritable bowel syndrome by carrying out gastrointestinal tests and questionnaires.

Understanding how diet and fiber affect GI function potentially will benefit the large numbers of children with irritable bowel syndrome (IBS) and provide insight into prevention of IBS in at risk children. We expect that the results from these studies can be used to lessen significantly the huge financial burden to society caused by these chronic conditions.

Consent will be obtained from the parent/guardian and assent from the child.

DETAILED DESCRIPTION:
Children with recurrent abdominal pain (RAP) who meet the criteria for irritable bowel syndrome (IBS) will be recruited and studied. They will have been diagnosed by a pediatric gastroenterologist and will have had at least one healthcare visits in the past year for the complaint of abdominal pain.

Coordinators will come out to the family's home on an evening that is convenient. Both the parent and child will fill out some questionnaires. Next, the parent and child will get instructions on how to fill out a diary to record any stomach pain the child is having and what their stools look like. The child will also collect a stool sample during the regular diet and diary collection period. Once the child has completed the diary, the child will go on a special diet for eight days to remove foods that may cause stomach pain (foods and drinks containing lactose, fructose, and sorbitol will be eliminated).

Two weeks later, the coordinators will come out to the family's home again to review the pain and stool diary that the child kept while on the special diet. The coordinators will explain how to collect some samples of urine, stool, and breath. These tests will evaluate the gastrointestinal (GI) tract for inflammation and transit time. If the special diet does not make the stomach pain go away, the child will be selected at random, like the flip of a coin, to be placed in one of two groups: one group that receives fiber or one group that receives a placebo or sugar pill. Fiber has been suggested to help children with stomach pain.

After the child has been on the treatment for 6 weeks, he/she will keep another diary and collect another set of samples of urine, stool, and breath.

The children will be followed at 3 months, 6 months and 18 months after the treatment period.

Children will be asked to collect additional stools

ELIGIBILITY:
Inclusion Criteria:

* Children who have had at least one physician visit in the past year for abdominal pain or IBS symptoms.
* Children with recurrent abdominal pain who meet the criteria for irritable bowel syndrome.

Exclusion Criteria:

* Children who have another disease that accounts for stomach pain
* Current use of anti-inflammatory medication
* Children taking a GI medication that makes pain go away completely
* Children with other chronic conditions including chronic pain conditions (e.g. heart condition, diabetes)
* Children who have decreased growth
* GI blood loss
* Unexplained fever
* Chronic severe diarrhea
* Weight loss of > or = to 5% of body weight within 3 month prior to enrollment
* History of abdominal surgeries
* A history of suicide
* Cognitive impairment significantly below average age and/or grade level
* Non-English speaking parent or child
* Vomiting >2x/month
* Children currently in psychotherapy for abdominal pain.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2009-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Improvement in pain and stooling symptoms | The last two weeks of treatment and up to 18 months after treatment

SECONDARY OUTCOMES:
Child anxiety, somatization, and coping | Four weeks prior to treatment and 6 months after treatment
Parental somatization, coping, and illness interaction | Four weeks prior to treatment and 6 months after treatment
Changes in GI Transit time | Prior to and after treatment
Changes in Breath Hydrogen production | Prior to and after treatment
Changes in GI Permeability | Prior to and after treatment
Changes in fecal calprotectin concentration | Prior to and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shulman, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Background] Shulman RJ, Eakin MN, Jarrett M, Czyzewski DI, Zeltzer LK. Characteristics of pain and stooling in children with recurrent abdominal pain. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):203-8. doi: 10.1097/01.mpg.0000243437.39710.c0. PMID 17255832
- [Background] Thakkar K, Gilger MA, Shulman RJ, El Serag HB. EGD in children with abdominal pain: a systematic review. Am J Gastroenterol. 2007 Mar;102(3):654-61. doi: 10.1111/j.1572-0241.2007.01051.x. PMID 17222318
- [Background] Czyzewski DI, Eakin MN, Lane MM, Jarrett M, Shulman RJ, M D. Recurrent Abdominal Pain in Primary and Tertiary Care: Differences and Similarities. Child Health Care. 2007 May 2;36(2):137-153. doi: 10.1080/02739610701334970. No abstract available. PMID 20357915
- [Background] Jarrett M, Heitkemper M, Czyzewski DI, Shulman R. Recurrent abdominal pain in children: forerunner to adult irritable bowel syndrome? J Spec Pediatr Nurs. 2003 Jul-Sep;8(3):81-9. doi: 10.1111/j.1088-145x.2003.00081.x. PMID 12942886
- [Background] Burr RL, Motzer SA, Chen W, Cowan MJ, Shulman RJ, Heitkemper MM. Heart rate variability and 24-hour minimum heart rate. Biol Res Nurs. 2006 Apr;7(4):256-67. doi: 10.1177/1099800405285268. PMID 16581896
- [Background] McOmber ME, Shulman RJ. Recurrent abdominal pain and irritable bowel syndrome in children. Curr Opin Pediatr. 2007 Oct;19(5):581-5. doi: 10.1097/MOP.0b013e3282bf6ddc. PMID 17885479
- [Background] Kellermayer R, Tatevian N, Klish W, Shulman RJ. Steroid responsive eosinophilic gastric outlet obstruction in a child. World J Gastroenterol. 2008 Apr 14;14(14):2270-1. doi: 10.3748/wjg.14.2270. PMID 18407608
- [Background] Amaizu N, Shulman R, Schanler R, Lau C. Maturation of oral feeding skills in preterm infants. Acta Paediatr. 2008 Jan;97(1):61-7. doi: 10.1111/j.1651-2227.2007.00548.x. Epub 2007 Dec 3. PMID 18052999
- [Background] McOmber MA, Shulman RJ. Pediatric functional gastrointestinal disorders. Nutr Clin Pract. 2008 Jun-Jul;23(3):268-74. doi: 10.1177/0884533608318671. PMID 18595859
- [Background] Shulman RJ, Eakin MN, Czyzewski DI, Jarrett M, Ou CN. Increased gastrointestinal permeability and gut inflammation in children with functional abdominal pain and irritable bowel syndrome. J Pediatr. 2008 Nov;153(5):646-50. doi: 10.1016/j.jpeds.2008.04.062. Epub 2008 Jun 9. PMID 18538790
- [Background] Lane MM, Weidler EM, Czyzewski DI, Shulman RJ. Pain symptoms and stooling patterns do not drive diagnostic costs for children with functional abdominal pain and irritable bowel syndrome in primary or tertiary care. Pediatrics. 2009 Mar;123(3):758-64. doi: 10.1542/peds.2008-0227. PMID 19254999
- [Derived] So SY, Badu S, Wu Q, Yalcinkaya N, Mirabile Y, Castaneda R, Musaad S, Heitkemper M, Savidge TC, Shulman RJ. Sex-Dependent Efficacy of Dietary Fiber in Pediatric Functional Abdominal Pain. Gastroenterology. 2024 Apr;166(4):645-657.e14. doi: 10.1053/j.gastro.2023.12.011. Epub 2023 Dec 19. PMID 38123024
- [Derived] Shulman RJ, Hollister EB, Cain K, Czyzewski DI, Self MM, Weidler EM, Devaraj S, Luna RA, Versalovic J, Heitkemper M. Psyllium Fiber Reduces Abdominal Pain in Children With Irritable Bowel Syndrome in a Randomized, Double-Blind Trial. Clin Gastroenterol Hepatol. 2017 May;15(5):712-719.e4. doi: 10.1016/j.cgh.2016.03.045. Epub 2016 Apr 11. PMID 27080737
- See also: Information about Kids GI Health — http://www.aboutkidsgi.org/
- See also: Information about Children in Clinical Research — http://www.childrenandclinicalstudies.nhlbi.nih.gov
- See also: Our research group's website at Baylor College of Medicine — http://www.bcm.edu/cnrc/kidsabdominalpain